CLINICAL TRIAL: NCT01567150
Title: Wound Fluid Protease Levels During Use of Novel Wound Dressing
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hollister Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5064-W
Record Dates: First submitted 2012-03-23; First posted 2012-03-30 (Estimated); Results first posted 2016-11-25 (Estimated); Last update posted 2016-11-25 (Estimated); Status verified 2016-10

CONDITIONS: Venous Stasis Ulcers
MeSH Terms: conditions — Varicose Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- novel dressing (Active Comparator): Treatment with novel dressing
  Interventions: Device: Novel Dressing
- Control (No Intervention): Control is treatment without novel dressing

INTERVENTIONS:
Device: Novel Dressing — Topical wound dressing
  Arms: novel dressing

SUMMARY:
This study is being conducted to characterize the way leg wounds respond to a new type of wound dressing, compared to wounds in patients who are not using the new dressing. The investigators will collect wound fluid for biochemical analysis, and they will measure the wound healing that occurs with and without the new dressing.

DETAILED DESCRIPTION:
Abnormal wound healing is characterized by prolonged inflammation and excess degradation of the extracellular matrix through the activity of proteinases and other enzymes. Wound fluids can provide biochemical information about the healing status of chronic wounds and the effects of wound treatments. In this study the investigators will obtain samples of wound fluid and measure healing in wounds randomized to receive the novel dressing or a control. The findings will be compared between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of venous insufficiency
* One or more partial or full-thickness venous leg ulcers 5-24 sq. cm in size without evidence of clinical infection
* Ankle/brachial index 0.8 and above
* Duration of wound up to one year
* Able to return to wound clinic for weekly evaluations
* Has signed Institutional Review Board approved informed consent

Exclusion Criteria:

* Exposed bone or tendon or necrotic wound base
* Signs or symptoms of cellulitis or osteomyelitis at the target ulcer
* Allergy to a component of the novel dressing or compression wrap
* Third degree burn
* Vasculitis, severe rheumatoid arthritis or other collagen vascular disease
* Receiving antibiotics
* Pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2012-02; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ginger Salvadalena, PhD, RN, Study Director — Hollister Incorporated
Locations (8):
- United States (8):
  - Arizona Heart Hospital, Phoenix, Arizona
  - Phoenix Baptist Hospital, Phoenix, Arizona
  - University of Miami, Department of Surgery, Div. of Vascular Surgery, Miami, Florida
  - Alexian Brothers Medical Center Wound Healing Center, Elk Grove Village, Illinois
  - Genesys Regional Medical Center, Grand Blanc, Michigan
  - NYU Langone Medical Center, New York, New York
  - Circleville Foot & Ankle, Circleville, Ohio
  - Baylor University Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 4 subjects attended only one study visit thus did not have evaluable data
Period: Overall Study
Arm/Group | Novel Dressing | Control
Started | 21 | 18
Completed | 19 | 16
Not Completed | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Novel Dressing | Control | Total
Number analyzed (Participants) | 19 | 16 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.1 (14.9) | 60.6 (12.9) | 58.1 (14.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 14
  Male | 12 | 9 | 21

OUTCOME MEASURES:

1. Primary Outcome: Matrix Metalloproteinase Level in Wound Fluid
Description: Wound fluid will be collected and analyzed at baseline and approximately every 7 days.
  Mean was calculated for each subject. Means and standard deviation were calculated for the treatment and control groups.
Time Frame: 8 weeks
Population: Overall mean across 8 week timeframe
Measure: Mean (Standard Deviation); unit: mcg/ml
Arm/Group | Novel Dressing | Control
Number analyzed (Participants) | 19 | 16
mcg/ml | 0.71 (0.78) | 0.88 (0.85)

2. Secondary Outcome: Wound Healing
Description: change in wound area mean was calculated for each subject Mean and sd were calculated for each group
Time Frame: 12 weeks
Population: average across 12 week time frame
Measure: Mean (Standard Deviation); unit: square cm
Arm/Group | Novel Dressing | Control
Number analyzed (Participants) | 19 | 16
square cm | -4.99 (8.22) | -2.49 (6.45)

ADVERSE EVENTS:
Time Frame: Up to 12 weeks
Arm/Group | Novel Dressing | Control
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/16
Other Adverse Events (participants affected / at risk) | 0/19 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less